CLINICAL TRIAL: NCT03429114
Title: Neural Correlates of Emotion Regulation and Executive Function in Binge Eating and Purging Among Adolescents
Brief Title: Emotion Regulation in Binge Eating and Purging Among Adolescents
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cara Bohon, PhD, Assistant Professo, Stanford University
Other Study IDs: 40075
Record Dates: First submitted 2018-02-02; First posted 2018-02-12 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Binge Eating; Purging (Eating Disorders)
MeSH Terms: conditions — Bulimia; Feeding and Eating Disorders | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Binge eating/purging: Adolescents engaging in recurrent binge eating and/or purging behavior.
  Interventions: Other: Magnetic resonance imaging
- Healthy comparison: Adolescents who do not have a history of eating disorders
  Interventions: Other: Magnetic resonance imaging

INTERVENTIONS:
Other: Magnetic resonance imaging — We will conduct MRI and fMRI brain scans to compare brain function between groups.

SUMMARY:
The study will examine the neural and behavioral correlates of emotion regulation in adolescents engaging in binge eating and/or purging and healthy adolescents. Furthermore, it will look at the influence of executive function on emotion regulation in this population. This study will allow us to gain further understanding of the neural basis of emotion regulation in this age group. Moreover, this study supports the need to develop new treatment approaches based on a better understanding of the brain processes associated with eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 14-18
* with or without current binge eating and/or purging behaviors

Exclusion Criteria:

We exclude patients of clinically significant low weight (<85% ideal body weight using CDC norms for height, age, and gender) and those with contraindications for MRI (e.g., orthodontia, metallic implants). Participants also will be without evidence of current or past major neurological (e.g., seizures, psychosis, head trauma) or major sensory deficit.

Ages: 14 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Female adolescents between ages 14-18.
Sampling Method: Non-Probability Sample
Enrollment: 47 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Brain activity during emotion conflict | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity during a task where participants respond to images of faces with emotional expressions overlaid with an emotion word written in text. We will focus on brain response during this task when emotion face vs word are in conflict.
Brain activity during emotion regulation | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity during a task where participants attempt to regulate emotional responses.
Brain activity during cognitive control and emotion response | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity during a task where participants engage in cognitive control and respond to emotional stimuli.

SECONDARY OUTCOMES:
Behavioral performance on emotion conflict task | Baseline
  Response times will be used as behavioral measure on the emotion conflict task
Behavioral performance on emotion regulation task | Baseline
  Emotion ratings will be used as behavioral measure on the emotion regulation task
Behavioral performance on cognitive control and emotion regulation task | Baseline
  Emotion ratings will be used as behavioral measure on the cognitive control and emotion regulation task

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Department of Psychiatry, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No